CLINICAL TRIAL: NCT06998706
Title: REGEND001 Autologous Basal Layer Stem Cell Transplantation for Interstitial Lung Disease (ILD): A Translational Application Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250515
Record Dates: First submitted 2025-05-15; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Lung Disease (ILD)
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICD patients (Experimental)
  Interventions: Biological: REGEND001 Autologous Basal Layer Stem Cell Suspension

INTERVENTIONS:
Biological: REGEND001 Autologous Basal Layer Stem Cell Suspension — REGEND001 Autologous Basal Layer Stem Cell Suspension is an innovative cell therapy product designed for chronic structural lung diseases, such as bronchiectasis. This treatment involves harvesting regenerative stem cells (expressing KRT5/P63 markers) from the patient's own bronchial basal layer via fiberoptic bronchoscopy. After isolation, purification, and ex vivo expansion, the cells are administered as a suspension through bronchoscopic infusion into damaged lung segments.

SUMMARY:
This clinical trial evaluates the safety and efficacy of REGEND001, an autologous bronchial basal layer stem cell therapy, in patients with interstitial lung disease (ILD). The treatment involves harvesting the patient's own stem cells (expressing KRT5/P63 markers), expanding them ex vivo, and administering them via bronchoscopic infusion to regenerate damaged lung tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years.
2. Confirmed diagnosis of ILD (e.g., IPF, connective tissue disease-associated ILD).
3. DLCO ≥30% and <80% predicted.

Exclusion Criteria:

1. Pregnancy, lactation, or plans for pregnancy within 1 year.
2. Active malignancy or history of malignancy.
3. Positive serology for HIV, HBV, HCV, or syphilis.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in DLCO from baseline. | Baseline, 4 weeks post treatment, 24 weeks post treatment
  The diffusing capacity of the lungs for carbon monoxide (DLCO) is a measurement of the gas transfer capacity of lung.

SECONDARY OUTCOMES:
Change in FVC from baseline | Baseline, 4 weeks post treatment, 24 weeks post treatment
  The forced vital capacity (FVC) is a measurement of the airflow capacity.
Incidence of adverse events and serious adverse events. | Through study completion, an average of 6 months
High-resolution CT (HRCT) imaging scores | Baseline, 4 weeks post treatment, 24 weeks post treatment
Quality of life (QoL) assessment via validated respiratory questionnaires | Baseline, 4 weeks post treatment, 24 weeks post treatment
  Score range: 0 to 100. Higher scores indicate a worse outcome

IPD SHARING:
Plan to Share IPD: No